CLINICAL TRIAL: NCT00545753
Title: A Phase 3 Comparative Safety and Efficacy Study Between NatrOVA Creme Rinse - 1% and NIX Creme Rinse in Subjects >6 Months of Age or Older With Pediculosis Capitis
Brief Title: Safety and Efficacy Study of NatrOVA Creme Rinse - 1% and NIX Creme Rinse in Subjects 6 Months or Older With Head Lice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPN-301-07
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Pediculosis
Keywords: Human Head lice
MeSH Terms: conditions — Lice Infestations | interventions — spinosad; Suspensions

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A - NatrOVA 1% - no nit combing (Experimental): NatrOVA Creme Rinse (spinosad) 1% - no nit combing required
  Interventions: Drug: Spinosad
- B - NatrOVA 1% - nit combing required (Experimental): NatrOVA Creme Rinse (spinosad) 1% - nit combing regimen required
  Interventions: Drug: Spinosad
- C - NIX (Active Comparator): NIX Creme Rinse (permethrin 1%) applied to Over the Counter (OTC) Instructions for Use
  Interventions: Drug: Permethrin 1%

INTERVENTIONS:
Drug: Spinosad — 10 minute topical application product, following by a complete rinse off.
  Other Names: Natroba (spinosad) Topical Suspension, 0.9%
  Arms: A - NatrOVA 1% - no nit combing
Drug: Spinosad — 10 minute topical application followed by a complete rinse off, followed by a nit combing regimen
  Other Names: Natroba (spinosad) Topical Suspension, 0.9%
  Arms: B - NatrOVA 1% - nit combing required
Drug: Permethrin 1% — Topical application for 10 minutes, followed by a complete rinse off, followed by a nit combing regimen
  Other Names: NIX Creme Rinse
  Arms: C - NIX

SUMMARY:
A comparative safety and efficacy study of NatrOVA Creme Rinse - 1% versus NIX Creme Rinse, under actual use conditions in subjects 6 months of age or greater who are infested with Pediculosis capitis (human head lice).

DETAILED DESCRIPTION:
This is a Phase 3 multi-site, randomized, evaluator/investigator-blinded, three-arm, parallel group study evaluating the safety and efficacy of NatrOVA Creme Rinse - 1% (with nit combing and without nit combing) versus NIX Creme Rinse in an "actual use" environment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have an active head lice infestation present at Day 0.
2. Subjects can be female or male, at least 6 months of age.
3. Subjects must be in good general health based on medical history.
4. Each subject must have an appropriately signed Informed Consent agreement. Subjects under the age of 12 must also provide written or oral assent.
5. The subject/caregiver must be able to read English or Spanish at a 7th grade level.
6. The parent or guardian within a household must be willing to allow other household members to be screened for head lice. If other household members are found to have a head lice infestation, they should also be enrolled in the study.
7. Subjects must agree to not use any other form of lice treatment during the course of the study and must agree not to use any of the excluded concomitant medications.
8. Subjects must agree not to cut or chemically treat their hair in the period between the initial treatment and the final visit.
9. Subjects/caregiver must demonstrate a clear understanding of his/her requirements for study participation and agree to comply with study instructions.

Exclusion Criteria:

1. Individuals with history of irritation or sensitivity to pediculicides or hair care products.
2. Individuals with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel or Sponsor, will interfere with the evaluation.
3. Individuals who require treatment with topical salicylic acid, topical corticosteroids, anthralin, vitamin D analogs, retinoids, immunosuppressants, topical hair growth formulations, and topical dandruff treatments.
4. Infested subjects who have been previously treated with a pediculicide within the 48 hours prior to the study.
5. Individuals with a condition or illness that, in the opinion of the Investigator, may compromise the objective of the protocol.
6. Individuals receiving systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel or study monitor may interfere with the study results.
7. Individuals who have participated in a clinical trial within the past 30 days.
8. Individuals (or individuals from households) who, in the opinion of the Investigator, do not understand the requirements for study participation and/or may be likely to exhibit poor compliance.
9. Individuals with household members who are infested with lice but are unwilling or unable to enroll in the study or to use the standard course of lice treatment.
10. Females who are pregnant or nursing. Females of childbearing potential must have a negative urine pregnancy test prior to treatment at Day 0. If a household has a pregnant female with an active case of head lice, the entire household is excluded from participation. If the pregnant household member does not have lice, this individual must NOT be the caregiver (one who provides treatment to other household members).
11. Sexually active females not using effective contraception.
12. Individuals who have a history of drug abuse in the past year.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bill Miller, MD, Study Director — Concentrics Research
Locations (6):
- United States (6):
  - Hill Top Research, Scottsdale, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Impact Clinical Trials, Beverly Hills, California
  - DMI Healthcare Group, Largo, Florida
  - Hill Top Research, Miamiville, Ohio
  - Haber Dermatology & Cosmetic Surgery, South Euclid, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject signed an informed consent and enrolled into the study on 25 September 2007; the last follow-up visit occurred on 22 April 2008.
Pre-assignment Details: After admission to the study, subjects could have withdrawn at any time for any reason such as they no longer met the eligibility criteria, personal reasons, etc.
Groups:
- A - NatrOVA 1% - No Nit Combing Required: NatrOVA Creme Rinse (spinosad) 1% - no nit combing required
- B - NatrOVA 1% - Nit Combing Required: NatrOVA Creme Rinse (spinosad) 1% - nit comb regimen required
- C - NIX Applied Per Over the Counter (OTC) Instructions: NIX Creme Rinse (permethrin 1%) applied to Over the Counter (OTC) Instructions for Use
Period: Overall Study
Arm/Group | A - NatrOVA 1% - No Nit Combing Required | B - NatrOVA 1% - Nit Combing Required | C - NIX Applied Per Over the Counter (OTC) Instructions
Started | 243 | 59 | 256
Completed | 227 | 54 | 230
Not Completed | 16 | 5 | 26
Not completed — Withdrawal by Subject | 0 | 1 | 10
Not completed — Lost to Follow-up | 13 | 3 | 12
Not completed — Protocol Violation | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- A - NatrOVA 1% - No Nit Combing Required: NatrOVA Creme Rinse - 1% - no nit combing required
- B - NatrOVA 1% - Nit Combing Required: NatrOVA Creme Rinse - 1% - nit comb regimen required
- C - NIX Applied Per Over the Counter (OTC) Instructions: NIX Creme Rinse applied to Over the Counter (OTC) Instructions for Use
- Total: Total of all reporting groups
Arm/Group | A - NatrOVA 1% - No Nit Combing Required | B - NatrOVA 1% - Nit Combing Required | C - NIX Applied Per Over the Counter (OTC) Instructions | Total
Number analyzed (Participants) | 243 | 59 | 256 | 558
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 172 | 40 | 177 | 389
  Between 18 and 65 years | 70 | 19 | 78 | 167
  >=65 years | 1 | 0 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 16 (15) | 19 (16) | 17 (14) | 17 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 47 | 210 | 457
  Male | 43 | 12 | 46 | 101
Region of Enrollment [Number; unit: participants]
  United States | 243 | 59 | 256 | 558

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of NatrOVA Creme Rinse - 1% Relative to NIX Creme Rinse in Subjects Infested With Head Lice
Description: The primary efficacy endpoint was the proportion of primary subjects in the enrolled households who were lice free (no live lice, adults or nymphs), as assessed by the trained evaluator, 14 days after the last treatment (i.e., Day 14 for subjects who treated once and Day 21 for subjects who treated twice).
Time Frame: Assessment were made 14 days following the final product treatment
Population: Primary efficacy analysis was conducted using the Intent to Treat data obtained from primary subjects (i.e., youngest enrolled members of each household who had at least three live lice at the time of entry into the study). Subjects who were lice free 14 days post-treatment were considered successes and all other subjects were considered failures.
Measure: Number; unit: participants
Groups:
- C - NIX Applied Per Over the Counter (OTC) Instructions: NIX Creme Rinse (permethrin 1%) applied according to Over the Counter (OTC)Instructions for Use
Arm/Group | A - NatrOVA 1% - No Nit Combing Required | B - NatrOVA 1% - Nit Combing Required | C - NIX Applied Per Over the Counter (OTC) Instructions
Number analyzed (Participants) | 91 | 23 | 89
participants
  Success (no live lice present) | 77 | 19 | 40 [32.7% to 57.5%]
  Failure (live lice present) | 14 | 4 | 49

2. Secondary Outcome: Evaluation of the Safety of NatrOVA Creme Rinse - 1% Based Upon Reported Adverse Events and Observed Skin/Scalp Reactions.
Description: To evaluate the safety of NatrOVA® 1% Creme Rinse based upon reported adverse events and observed skin/scalp reactions. Additional safety assessments included cutaneous/ocular irritation.
Time Frame: Participants were followed for a minimum of 14 days (1 treatment) and a maximum of 21 days (2 treatments)
Population: 558 subjects were randomized to treatment and 540 subjects used the study drug and returned for at least one post-baseline evaluation. At Day 0 the study drug was to be used within 24 hours. At Day 7 if subject presented with live lice they were provided a second treatment to be used within 24 hours. Thus subjects used 1 or 2 treatments.
Measure: Number; unit: Incidents
Groups:
- A/B - NatrOVA 1% - With/Without Nit Combing: NatrOVA Creme Rinse (spinosad) 1% - With or without nit combing required
Arm/Group | A/B - NatrOVA 1% - With/Without Nit Combing | C - NIX Applied Per Over the Counter (OTC) Instructions
Number analyzed (Participants) | 294 | 246
Incidents
  Ear and labyrinth disorders - Ear pain | 0 | 1
  Eye disorders - Eye irritation | 0 | 3
  Eye disorders - pruritus | 0 | 1
  Eye disorders - Lacrimination increased | 0 | 1
  Eye disorders - Occular hyperaemia | 12 | 15
  Gastrointestinal disorders - Diarrhea | 1 | 0
  Gastrointestinal disorders - Stomach discomfort | 1 | 0
  Gastrointestinal disorders - Vomiting | 1 | 0
  Administration site conditions - discoloration | 0 | 1
  Administration site conditions - Dryness | 1 | 0
  Administration site conditions - Erythema | 15 | 17
  Administration site conditions - Irritation | 5 | 6
  Administration site conditions - Scab | 0 | 1
  General Disorder - Pyrexia | 1 | 1
  Infections and infestations - Cellulitis | 0 | 1
  Infections and infestations - Influenza | 1 | 0
  Infections and infestations - Nasopharyngitis | 1 | 2
  Infections and infestations - Otitis media | 1 | 0
  Infections - Pharyngitis streptococal | 0 | 1
  Infections - Upper respiratory tract infection | 0 | 3
  Injury - Skin laceration | 1 | 0
  Nervous system disorders - Headache | 1 | 1
  Nervous system disorders - Syncope | 0 | 1
  Respiratory -Chronic obstructive pulmonary disease | 0 | 1
  Respiratory - Cough | 1 | 1
  Respiratory disorders - pharyngolaryngeal pain | 1 | 0
  Skin disorders - Alopecia | 1 | 0
  Skin disorders - Dry skin | 1 | 1
  Skin disorders - Erythema | 1 | 4

ADVERSE EVENTS:
Time Frame: Through out the study (7 months).
Description: Verbatim descriptions of Adverse Events (AE) were assigned to system organ classes and terms via the MedDRA dictionary (v10.1). All randomized subjects who were presumed to have used the study medication at least once and who provided at least one post-baseline evaluation or reported at least one AE subsequent to using the study medication.
Groups:
- A/B - NatrOVA 1% - With/Without Nit Combing: NatrOVA Creme Rinse - 1% - With or without nit combing
Arm/Group | A/B - NatrOVA 1% - With/Without Nit Combing | C - NIX Applied Per Over the Counter (OTC) Instructions
Serious Adverse Events (participants affected / at risk) | 0/294 | 2/246
Other Adverse Events (participants affected / at risk) | 34/294 | 49/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/B - NatrOVA 1% - With/Without Nit Combing (N=294) | C - NIX Applied Per Over the Counter (OTC) Instructions (N=246)
Application Site Erythema (General disorders) | 0 (0) | 1 (1) — Subject randomized to NIX, applied the study medication twice. Day 8 the subject presented with application site erythema. Investigator reported event as a serious AE despite the fact that it did not meet the regulatory definition of a serious event.
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Subject randomized to NIX, applied study medication twice. Day 14 presented with cellulitis. Subject was hospitalized, considered mild severity and unrelated to study medication. The event resolved with no sequelae. Subject didn't have Day 21 visit.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/B - NatrOVA 1% - With/Without Nit Combing (N=294) | C - NIX Applied Per Over the Counter (OTC) Instructions (N=246)
Eye irritation (Eye disorders) | 0 (0) | 3 (3)
Occular hyperaemia (Eye disorders) | 12 (12) | 15 (15)
Application site erythema (General disorders) | 15 (15) | 16 (16)
Application site irritation (General disorders) | 5 (5) | 6 (6)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No